CLINICAL TRIAL: NCT06677814
Title: Development and Validation of an Anxiety Disorder Prediction Model for Premature Ejaculation Patients
Status: Recruiting | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY 20212177-F-1
Record Dates: First submitted 2024-10-31; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-10

CONDITIONS: Premature Ejaculation; Anxiety
MeSH Terms: conditions — Premature Ejaculation; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training cohort: This cohort data will be used to screen for independent risk factors for anxiety disorders in patients with premature ejaculation and to initially construct a risk prediction model.
- Validation cohort: This cohort data will be used to verify the performance and stability of the risk prediction model to ensure the promotion and use of the model.

SUMMARY:
Background:

Premature ejaculation (PE) is a common sexual dysfunction that can significantly impact the quality of life and psychological well-being of affected individuals. Anxiety disorders, often comorbid with PE, exacerbate symptoms and complicate treatment outcomes. There is a critical need for a reliable prediction model to identify patients at risk of developing anxiety disorders associated with PE.

Objective:

The primary aim of this study is to develop and validate a predictive model that accurately identifies premature ejaculation patients who are at high risk of developing anxiety disorders. The model will be designed to facilitate early intervention strategies and improve patient outcomes.

Methods:

This prospective observational study will enroll male patients diagnosed with PE from multiple clinical centers. Participants will undergo comprehensive assessments including validated questionnaires, clinical interviews, and medical history reviews to collect baseline data on potential predictors of anxiety disorders. Machine learning algorithms will be utilized to analyze the collected data and derive a predictive model. External validation will be conducted using a separate cohort of patients not involved in the initial model development phase.

Outcome Measures:

The primary outcome measure will be the accuracy of the predictive model in identifying patients who subsequently develop anxiety disorders within a predefined follow-up period. Secondary outcomes include evaluating the model's sensitivity, specificity, positive predictive value, and negative predictive value.

Significance:

Successful development and validation of this prediction model could lead to improved patient care through targeted interventions and personalized treatment plans for those at risk of anxiety disorders related to PE. This research may also contribute to a better understanding of the complex interplay between sexual dysfunction and mental health.

ELIGIBILITY:
Inclusion Criteria:

* Comply with the international medical premature ejaculation diagnostic criteria
* Individuals with a "heterosexual" orientation who engage in vaginal intercourse
* Having a stable relationship with "monogamy"
* The International Index of Erectile Function-5 scale is ≥17 points, indicating that the patient has no erectile dysfunction or only mild erectile dysfunction
* Be informed of the purpose of this study, support this study, and complete the informed consent form

Exclusion Criteria:

* Minors under the age of 18
* Individuals with a sexual orientation of "gay" or "bisexual"
* The judgment of "ejaculation too fast" is based only on masturbation or non-vaginal sexual intercourse
* The score of the premature ejaculation self-assessment scale is ≤8 points
* Suffering from diseases that may affect anxiety symptoms (hyperthyroidism/hypothyroidism, digestive diseases, malignant tumors, etc.)
* Within 2 months, have taken anti-anxiety drugs and/or drugs for PE treatment
* Those with a history of severe neurological diseases (such as epilepsy) and/or a history of schizophrenia, bipolar disorder, or other mental disorders
* Poor cooperation during diagnostic interviews

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants for this study will be male patients diagnosed with premature ejaculation (PE).
  Sample Size： Approximately 700 patients are expected to be recruited for this study. The sample size was determined based on previous studies and statistical calculations to ensure adequate statistical power.
  Recruitment Sites： Participants will be recruited from four tertiary hospitals within the country.
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-03-25 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Anxiety State of patients | Within three months after the patient is diagnosed with premature ejaculation.
  Use the Mini International Neuropsychiatric Interview (MINI) to conduct a structured interview with the patient to determine if they have an anxiety disorder.
Accuracy of the Prediction Model | Through study completion, an average fo 1 year
  Evaluate the accuracy of the prediction model by comparing its predictions against actual diagnoses of anxiety disorders.

SECONDARY OUTCOMES:
Sensitivity of the Prediction Model | Through study completion, an average fo 1 year
  Assess the model's performance in identifying patients who actually develop anxiety disorders.
Specificity of the Prediction Model | Through study completion, an average fo 1 year
  Assess the model's performance in identifying patients who do not develop anxiety disorders.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Xi'an Daxing Hospital affiliated to Yan'an University, Xi'an, Shaanxi
  - Xijing Hospital, Xi'an, Shaanxi